CLINICAL TRIAL: NCT06212258
Title: Pneumoperitoneum Increases Mean Expiratory Flow Rate: an Observational Study in Healthy-lung Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Balázs Sütő (Other)
Responsible Party: Sponsor-Investigator, Balázs Sütő, Consultant Anaesthetist, University of Pecs
Organization: University of Pecs (Other)
Other Study IDs: 9746 - PTE - 2023
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Pneumoperitoneum Increases Mean Expiratory Flow Rate
Keywords: mechanical ventilation; body mass index; chest compliance; pneumoperitoneum; expiratory flow rate, intraabdominal pressure, laparoscopic surgery
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Abdominal Laparascopy — pneumoperitoneum

SUMMARY:
Upon introducing pneumoperitoneum our research team noticed a reduction in expiration time displayed on the screen of the anesthesia machine. Since most respirators do not directly indicate the length of expiratory time and the average expiratory flow rate, we decided to investigate whether pneumoperitoneum really accelerates expiratory flow rate and thus shortens expiratory time.

DETAILED DESCRIPTION:
Furthermore we also intended to investigate which ventilation parameters these changes can be correlated with, elucidating the factors contributing to the acceleration of expiration..

This study aims to uncover the physiological mechanisms behind alterations in respiratory dynamics during and after pneumoperitoneum, offering valuable insights that may aid in refining ventilation strategies in the context of laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic abdominal surgery, healthy lung patients, age over 18 years. Obrained, written informed consent to partake in the research.

Exclusion Criteria:

chronic obstructive pulmonary disease, bronchial asthma, silicosis, and those with a history of previous lung surgery, patients under 18 years of age, those who had not provided consent, and pregnant individuals were excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Helthy lung patients, over age 18 years, males and femailes together.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Pneumoperitoneum increases mean expiratory flow rate | during surgery
  Elevated intraabdominal pressure leads to a decrease in respiratory compliance and an increase in peak inspiratory pressure., therefore (consequently), expiration commences with a higher pressure difference.
Expiration time would be shortened, resulting in a potentially higher flow rate | during surgery
  We assumed (hypothesized) that the expiration time would be shortened, resulting in a potentially higher flow rate compared to pre-pneumoperitoneum conditions. Additionally, we also conducted calculations to establish correlations between respiratory parameters and the mean increment in expiratory flow rate relative to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia and Intensive Care, Medical School, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided